CLINICAL TRIAL: NCT00241956
Title: Impact of Diabetes and Glucose Control During Rehabilitation After Stroke
Status: Terminated | Type: Observational
Why Stopped: poor data collection
Sponsor: Melbourne Health (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Dr Leo Rando, Royal Melbourne Hospital
Other Study IDs: 2004.246
Record Dates: First submitted 2005-10-18; First posted 2005-10-19 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: Cerebrovascular Accident; Diabetes; Hyperglycemia
MeSH Terms: conditions — Stroke; Diabetes Mellitus; Hyperglycemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To assess whether patients with diabetes have less clinical improvement during inpatient rehabilitation than those without diabetes and whether hyperglycaemia during rehabilitation is an adverse prognostic indicator.

DETAILED DESCRIPTION:
Patients with diabetes have a higher mortality rate and more severe disability from stroke compared to those without diabetes. Those with hyperglycaemia tend to progress to a larger final stroke size. Diabetes and hyperglycaemia may affect the ability of the patient to clinically improve, independent of the degree of initial impairment. We will perform a retrospective review of medical records of stroke patients admitted to an inpatient rehabilitation unit. We will compare outcomes of changes in disability scales (FIM and Barthel) from admission to discharge, length of stay and hospital events between those with and without diabetes. Amongst those with diabetes, we will also assess whether those with higher mean blood glucose levels during their inpatient rehabilitation stay have worse outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient rehabilitation for acute stroke

Exclusion Criteria:

* Medical records unavailable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Stroke rehab patients
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2005-10; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leo Rando, MBBS FRACP, Principal Investigator — Melbourne Health
Locations (1):
- The Royal Melbourne Hospital, Melbourne, Victoria, Australia